CLINICAL TRIAL: NCT00400959
Title: Intracoronary Injection of CD133+ Autologous Hematopoietic Cells After Myocardial Infarction
Brief Title: CD133+ Autologous Cells After Myocardial Infarction
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CFT92002
Record Dates: First submitted 2006-11-14; First posted 2006-11-17 (Estimated); Last update posted 2006-11-17 (Estimated); Status verified 2006-11

CONDITIONS: Acute Myocardial Infarction
Keywords: cell therapy; acute myocardial infarction

INTERVENTIONS:
Procedure: cd133+cell intracoronary administration

SUMMARY:
TITLE Intracoronary injection of CD133+ autologous hematopoietic cells after myocardial infarction.

TRIAL DESIGN Pilot phase I/II parallel group study, with an untreated control group.

SPONSOR IRCCS Ospedale Maggiore Policlinico Milano INDICATION Acute myocardial infarction (AMI). TARGET POPULATION Patients (pts) with AMI treated with Primary Coronary Angioplasty (PTCA) with successful recanalization but unsuccessful reperfusion (myocardial blush (MB) grade 0 or 1 and less than 70% ST segment elevation resolution (STeR) (see Poli et al., Circulation, 2002).

OBJECTIVES Primary:

1. To evaluate the safety of intracoronary injection of CD133+ cells from autologous bone marrow (ABM) and mobilized peripheral blood (MPB) in the target population.
2. To evaluate the efficacy, of the selective injection of CD133+ cells from ABM and MPB in the culprit vessel of the target population, on regional and global contractile function and on perfusion and metabolism of the infarcted area, depending on cell dose and comparing to controls.

   Secondary:
3. To evaluate the disease-related morbility of the target population.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent;
* age: 18-65 years;
* large acute myocardial infarction (due to proximal occlusion of the left anterior descending or the right coronary artery) after successful primary PTCA carried out between the IV and the XXIV hour from the onset of AMI symptoms;
* signs of microvascular dysfunction in the infarcted area: absence of STeR and angiographic MB, graded according to the dye density score (see van't Hof et al., Circulation, 1998); life expectancy more than 6 months.

Exclusion Criteria:

* Pregnancy;
* indication to aorto-coronaric by-pass;
* neoplasia (previous or in progress);
* primary diseases of the BM;
* diabetes;
* immunosuppressive therapy;
* laboratory alterations of protein S, protein C, ATIII or Fibrinogen;
* severe co-morbidity.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15
Dates: Start 2004-06; Study Completion 2006-10

PRIMARY OUTCOMES:
myocardial flow (MF) (mL/g/min) evaluated by Positron Emission Tomography(PET) with Nitrogen-13 ammonia (13NH3),
Ejection fraction (%) evaluated by 2D echocardiography;

SECONDARY OUTCOMES:
perfusion/metabolism mismatch (P/Mm) evaluated by PET with Fluorine-18 fluorodeoxyglucose (FDG);
Left Ventricular Wall Motion Score Index (LVWMSI) evaluated by 2D

CONTACTS AND LOCATIONS:
Overall Officials: Rosaria Giordano, MD, Principal Investigator — Cell Factory Department of Regenerative Medicine Policlinic Milan
Locations (1):
- Cell Factory, department of regenerative medicine, Policlinic of Milan, Milan, Italy

REFERENCES:
- [Derived] Colombo A, Castellani M, Piccaluga E, Pusineri E, Palatresi S, Longari V, Canzi C, Sacchi E, Rossi E, Rech R, Gerundini P, Viecca M, Deliliers GL, Rebulla P, Soligo D, Giordano R. Myocardial blood flow and infarct size after CD133+ cell injection in large myocardial infarction with good recanalization and poor reperfusion: results from a randomized controlled trial. J Cardiovasc Med (Hagerstown). 2011 Apr;12(4):239-48. doi: 10.2459/JCM.0b013e328343d708. PMID 21372740